CLINICAL TRIAL: NCT06182397
Title: MAGICAL BTK: Randomized Controlled Trial of MAGIcTouch - Sirolimus Coated BALloon Versus Standard Balloon Angioplasty in The Treatment of Below The Knee Arterial Disease
Brief Title: Sirolimus Coated BALloon Versus Standard Balloon Angioplasty in The Treatment of Below The Knee Arterial Disease
Acronym: MAGICAL BTK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Concept Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CM-US-R04
Record Dates: First submitted 2023-12-04; First posted 2023-12-26 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Arterial Disease of Legs; Below-the-knee Obstruction; PAD - Peripheral Arterial Disease
Keywords: below the knee; PTA; Angioplasty; lower limb

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a single-blinded clinical investigation in which subjects will be blinded.The physician performing the index procedure will not be blinded. It is recommended, where feasible, that a different physician, or qualified designee, who is blinded to the subject's treatment, conduct protocol-required follow-up visits. The Study Coordinator will be unblinded.
  The technologists performing follow-up ultrasound scans, the Clinical Events Committee, the Data Safety Monitoring Board and core laboratories will be blinded. In emergency situations, the treating physician is responsible for assessing whether unblinding the treatment assignment is necessary, with the subject's safety as the first priority in making such a decision. If the treating physician decides that unblinding is warranted, the investigator will contact Concept Medical or the CRO to obtain the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- MagicTouch PTA sirolimus DCB (Active Comparator): MagicTouch PTA sirolimus drug coated balloon (DCB) in addition to standard balloon angioplasty
  Interventions: Device: MagicTouch PTA Sirolimus drug coated balloon
- Placebo balloon angioplasty (Placebo Comparator): Placebo balloon angioplasty in addition to standard balloon angioplasty (PTA)
  Interventions: Device: Placebo balloon angioplasty

INTERVENTIONS:
Device: MagicTouch PTA Sirolimus drug coated balloon — All patients must first be treated with pre dilatation with a standard balloon angioplasty using any standard balloon catheters at the discretion of the operator. Magic Touch PTA Sirolimus coated balloon catheter is an adjunct treatment that should be used in combination with standard balloon angioplasty. Following successful crossing of wire across the lesion and plain balloon angioplasty of arterial lesion with successful lesion preparation with residual lesion <30%, subjects will be randomized to receive study device balloon. If patients are assigned to MagicTouch PTA Sirolimus DCB, the Angioplasty of lower limb will be performed with this device in addition to standard balloon angioplasty.
  Arms: MagicTouch PTA sirolimus DCB
Device: Placebo balloon angioplasty — For participants randomized to a Placebo balloon angioplasty group, a Placebo balloon angioplasty in addition to standard balloon angioplasty will be performed.
  Arms: Placebo balloon angioplasty

SUMMARY:
This is a Pivotal, Prospective, randomized, two arm, placebo controlled, single-blind, multicenter trial that will be conducted at approximately 80 sites; approx. 50 sites with at least 50% of subjects will be recruited from USA and approx. 30 sites OUS - Europe, Australia and Asia. Each site will be capped at 30 maximum subjects recruited.

The main goal of this clinical trial is to determine the effectiveness and safety of the sirolimus drug coated balloon (DCB) versus standard percutaneous transluminal angioplasty (PTA) for the treatment of below the knee arterial disease.

Eligible subjects will be randomised in a 1:1 allocation ratio and stratified by recruiting countries. Each subject will be randomized to receive either:

1. MagicTouch PTA sirolimus coated balloon catheter (DCB) in addition to standard balloon angioplasty or
2. Placebo balloon angioplasty in addition to standard balloon angioplasty (PTA).

DETAILED DESCRIPTION:
The burden of limb loss because of peripheral arterial disease (PAD) is high and this problem is set to worsen globally. Treatment of PAD primarily involves revascularisation of the limb. Angioplasty as a first line strategy of revascularization over surgical procedures has been adopted by many vascular centres. In recent years, studies have shown that local drug delivery using drug coated balloons (DCB) during angioplasty for PAD can successfully deliver effective local tissue concentrations of antiproliferative drugs to the lesions in the artery involved in the PAD. This offers the potential for sustained anti-restenotic efficacy.

Randomized trials have shown superiority of Paclitaxel DCBs over just plain-balloon angioplasty for treatment of femoropopliteal occlusive disease, and DCB is now considered the standard of care in many regions. However, the efficacy of Paclitaxel below the knee is less clear, as multiple randomized trials evaluating Paclitaxel-coated DCBs below the knee have failed to meet their primary endpoints. Alternative drugs for DCBs are therefore needed and sirolimus may offer an attractive alternative. Compared to Paclitaxel, sirolimus is cytostatic in its mode of action with a high margin of safety. It has a high transfer rate to the vessel wall and has been shown to effectively inhibit neointimal hyperplasia in the porcine coronary model. In the coronary artery interventions, preliminary clinical studies using Sirolimus DCBs have also shown excellent procedural and 6- & 12- months patency. This study aims to conduct a single blind, randomised controlled multicentre trial of sirolimus drug coated balloon versus standard percutaneous transluminal angioplasty in patients with below the knee arterial disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 years or minimum age (is allowed the inclusion of subjects > 21 years OR adulthood minimum age (depending on the US state regulations)
2. Rutherford class 4 with documented WIFI score, not exceeding more than 30% of target patient population.
3. Rutherford class 5 to 6 in the target limb with documented WIFI score.

   Intraoperative Inclusion Criteria:
4. Single or sequential de novo or re-stenotic lesions (stenosis of > 50% or occlusions) from 2 to 20cm in the proximal 200mm of below the knee arteries. Lesion is considered as one lesion if there is maximum of 30 mm gap between lesions at discretion of investigator. Below the knee arteries are Tibio-peroneal trunk, Peroneal bifurcation, anterior tibial artery, posterior tibial artery and peroneal artery. With documented Distal Run off a maximum of two tibial vessels can be treated in the index procedure. Inflow free from flow limiting lesions (<50% stenosis) confirmed by duplex or angiography. Subjects with flow limiting inflow lesions (>50% stenosis) can be included if lesion had been treated successfully (<30% residual stenosis) before or during the index procedure.
5. Target vessel has angiographically documented unimpaired (<50% stenosis) run off into a named Tibio-pedal artery (Peroneal, Anterior Tibial/ Dorsalis Pedis/ Posterior Tibial Artery)

Exclusion Criteria:

1. Comorbid conditions limiting life expectancy ≤ 1 year
2. Subject is currently participating in another investigational drug or device study that has not reached first primary endpoint yet
3. Subject is lactating, pregnant or planning to become pregnant during the course of the study
4. Subject with extensive tissue loss salvageable only with complex foot reconstruction or non-traditional trans metatarsal amputation. This includes subjects with:

   1. Osteomyelitis including and/or proximal to the metatarsal head
   2. Gangrene involving the plantar skin of the forefoot, midfoot,or heel
   3. Deep ulcer or large shallow ulcer (> 3 cm) involving the plantar skin of the forefoot, midfoot, or heel
   4. Full thickness heel ulcer with/without calcaneal involvement
   5. Any wound with calcaneal bone involvement
   6. Wounds that are deemed to be neuropathic or non-ischemic in nature
   7. Wounds that would require flap coverage or complex wound management for large soft tissue defect
   8. Full thickness wounds on the dorsum of the foot with exposed tendon or bone
5. Prior bypass surgery of target vessel
6. Planned amputation of the target limb (major)
7. Previously implanted stent in the target lesion
8. Vulnerable or protected adults
9. Bleeding diathesis or another disorder (i.e. gastrointestinal ulceration,etc) which would prevent the use of mandated antiplatelet agents
10. Known allergy to sirolimus
11. Subjects with severe (Stage 4) renal disease, defined eGFR < 30.

    Intraoperative exclusion criteria:
12. Failure to successfully cross the target lesion with a guide wire
13. Target vessel has lesions extending beyond the ankle joint
14. Failure to obtain <30% residual stenosis prior to randomization
15. Lesions requiring treatment through retrograde access . Retrograde wire crossing is allowed but treatment must be performed from the antegrade approach.
16. Use of commercially available DCBs, bare metal stents, drug eluting stents, specialty balloons or atherectomy devices at the target lesions. (Non-compliant balloons are not considered specialty balloons). For Inflow and non-target lesions all the approved devices are allowed.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2031-02-01 (Estimated)

PRIMARY OUTCOMES:
Primary patency at 12 months defined as freedom from Target Vessel Occlusion, Binary Restenosis, Clinically-Driven Target Lesion Revascularization and Major Amputation. | 12 months
  Binary restenosis will be defined as the proportion of subjects with duplex ultrasonography-derived peak systolic velocity ratio of > 2.0 with correlating factors. If the PSV at the reference area in the vessel is abnormal, the core laboratory will employ the following other criteria to diagnose a stenosis of > 50%:
  * Monophasic/ low resistive waveforms (parvus tardus) at the stenotic area or distal to an acoustic shadow
  * Post-stenotic turbulence distal to the stenosis, along with a decrease in peak systolic velocities Gray scale/ B-mode imaging demonstrates significant plaque with stenosis along with a focal increase in the absolute PSV value.
  * Occlusion = Absence of color filling and spectral Doppler signal.
Composite safety endpoint | 6-months for n.1 and n.2; 30 days for n.3
  Proportion of subjects who experienced any of the following:
  1. 6-month above ankle major amputation of the index limb,
  2. 6-month major re-intervention (i.e., angioplasty of target lesion, new bypass graft, jump/interposition graft, or thrombectomy or thrombolysis)
  3. Perioperative (30 day) mortality.

SECONDARY OUTCOMES:
Secondary Safety endpoint 1 | 1, 6, 12, 24, 36, 48 and 60 months
  Proportion of device and procedure related death
Secondary Safety endpoint 2 | 1, 6, 12, 24, 36, 48 and 60 months
  Proportion of subjects with death by any cause
Secondary Safety endpoint 3 | 1, 6, 12, 24, 36, 48 and 60 months
  Proportion of subjects with major target limb amputation
Secondary Safety endpoint 4 | From day 0 to day 14
  Proportion of subjects with target vessel thrombosis
Secondary Safety endpoint 5 | From day 0 to 60 months
  Occurrence of adverse events (AEs), serious AEs and AEs related to device and procedure
Secondary efficacy endpoints 1 | From day 0 to 60 months
  Proportion of subjects with acute procedural success
Secondary efficacy endpoints 2 | 6, 12, 24, and 36 months
  Proportion of subjects who are free from clinically driven Target Lesion Revascularization (CD-TLR)
Secondary efficacy endpoints 3 | 6,12,24 and 36 months
  Proportion of subjects who are free from Target Vessel Revascularization (TVR)
Secondary efficacy endpoints 4 | 24 months
  Primary patency, defined as a composite of freedom from Target Vessel Occlusion, Binary Restenosis, Clinically Driven Target Lesion Revascularization and Major Amputation
Secondary efficacy endpoints 5 | 6, 12 and 24 months
  Proportion of subjects with restenosis. Restenosis is defined by duplex ultrasonography-derived peak systolic velocity ratio of >2.0 and <4.0
Secondary efficacy endpoints 6 | 6, 12, 24, 36, 48 and 60 months
  Amputation-free survival
Secondary efficacy endpoints 7 | 6,12, 24, 36, 48 and 60 months
  Proportion of subjects with clinical success defined as Improvement of ≥1 category in Rutherford classification compared to the pre-procedure Rutherford classification
Secondary efficacy endpoints 8 | From day 0 to day 1
  Proportion of subjects with technical success
Secondary efficacy endpoints 9 | 1, 3, 6, and 12 months
  Wound assessment. Follow-up will cease once wound completely heals as adjudicated by the core lab.
Secondary efficacy endpoints 10 | 6, 12 and 24 months
  Mean change from baseline in Toe pressure and ABI assessment
Secondary Functional endpoints 1 | 6,12, 24, and 36 months
  Mean change from baseline in EuroQol 5-dimension 5-level (EQ-5D-5L) health-related quality of life questionnaire's VAS score and utility index.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Secondary Functional endpoints 2 | 6,12, 24, and 36 months
  Mean change from baseline in walking impairment questionnaire score. In the WIQ distance score, the degree of difficulty in the walking of specific distances is ranked on a 0 to 4 Likert scale, in which 0 represents the inability to walk the distance and 4 represents no difficulty. A Likert scale is an ordinal scale of consecutive, equidistant, numerical values (ie, 0 to 4).

CONTACTS AND LOCATIONS:
Overall Officials: Sahil Parikh, MD, Study Chair — New York-Presbyterian/Columbia University Irving Pavilion
Locations (29):
- United States (29):
  - Honor Health Research & Innovation Institute, Scottsdale, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Vascular Institute of the Midwest, Davenport, Iowa
  - Unity Point Health Des Moines, Des Moines, Iowa
  - Atria Vascular and Vein, Farmington Hills, Michigan
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Virtua Healthcare - Virtua Our Lady of Lourdes, Marlton, New Jersey
  - Northwell Health Long Island Jewish Medical Center, Lake Success, New York
  - NYU Langone Medical Center, New York, New York
  - The Mount Sinai Hospital, New York, New York
  - Columbia University Irving Medical center/NYPH, New York, New York
  - New York Presbyterian - Weill Cornell Medical Center Vascular & Endovascular Surgery, New York, New York
  - St. Francis Hospital and Heart Center, Roslyn, New York
  - Westchester Medical Center, Valhalla, New York
  - The Christ Hospital Network Outpatient Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Lankenau Institute for Medical Research Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - University of Pennsylvania - Penn Heart and Vascular Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina(MUSC) Health Ashley River Tower, Charleston, South Carolina
  - Ascension Seton Medical Center Austin, Austin, Texas
  - Baylor Research Institute, Dallas, Texas
  - HOPE Vascular and Podiatry, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - San Antonio Vascular and Endovascular Clinic, San Antonio, Texas
  - University of Washington Seattle, Seattle, Washington

REFERENCES:
- [Result] Giacoppo D, Cassese S, Harada Y, Colleran R, Michel J, Fusaro M, Kastrati A, Byrne RA. Drug-Coated Balloon Versus Plain Balloon Angioplasty for the Treatment of Femoropopliteal Artery Disease: An Updated Systematic Review and Meta-Analysis of Randomized Clinical Trials. JACC Cardiovasc Interv. 2016 Aug 22;9(16):1731-42. doi: 10.1016/j.jcin.2016.06.008. PMID 27539695
- [Result] Clever YP, Peters D, Calisse J, Bettink S, Berg MC, Sperling C, Stoever M, Cremers B, Kelsch B, Bohm M, Speck U, Scheller B. Novel Sirolimus-Coated Balloon Catheter: In Vivo Evaluation in a Porcine Coronary Model. Circ Cardiovasc Interv. 2016 Apr;9(4):e003543. doi: 10.1161/CIRCINTERVENTIONS.115.003543. PMID 27069105
- [Result] Verheye S, Vrolix M, Kumsars I, Erglis A, Sondore D, Agostoni P, Cornelis K, Janssens L, Maeng M, Slagboom T, Amoroso G, Jensen LO, Granada JF, Stella P. The SABRE Trial (Sirolimus Angioplasty Balloon for Coronary In-Stent Restenosis): Angiographic Results and 1-Year Clinical Outcomes. JACC Cardiovasc Interv. 2017 Oct 23;10(20):2029-2037. doi: 10.1016/j.jcin.2017.06.021. Epub 2017 Sep 27. PMID 28964764
- [Result] Patel A, Irani FG, Pua U, Tay KH, Chong TT, Leong S, Chan ES, Tan GWL, Burgmans MC, Zhuang KD, Quek LHH, Kwan J, Damodharan K, Gogna A, Tan BP, Too CW, Chan SXJM, Chng SP, Yuan W, Tan BS. Randomized Controlled Trial Comparing Drug-coated Balloon Angioplasty versus Conventional Balloon Angioplasty for Treating Below-the-Knee Arteries in Critical Limb Ischemia: The SINGA-PACLI Trial. Radiology. 2021 Sep;300(3):715-724. doi: 10.1148/radiol.2021204294. Epub 2021 Jul 6. PMID 34227886
- [Result] Choke E, Tang TY, Peh E, Damodharan K, Cheng SC, Tay JS, Finn AV. MagicTouch PTA Sirolimus Coated Balloon for Femoropopliteal and Below the Knee Disease: Results From XTOSI Pilot Study Up To 12 Months. J Endovasc Ther. 2022 Oct;29(5):780-789. doi: 10.1177/15266028211064816. Epub 2021 Dec 15. PMID 34911383
- [Result] Rosenfield K, Jaff MR, White CJ, Rocha-Singh K, Mena-Hurtado C, Metzger DC, Brodmann M, Pilger E, Zeller T, Krishnan P, Gammon R, Muller-Hulsbeck S, Nehler MR, Benenati JF, Scheinert D; LEVANT 2 Investigators. Trial of a Paclitaxel-Coated Balloon for Femoropopliteal Artery Disease. N Engl J Med. 2015 Jul 9;373(2):145-53. doi: 10.1056/NEJMoa1406235. Epub 2015 Jun 24. PMID 26106946
- [Result] Steiner S, Willfort-Ehringer A, Sievert H, Geist V, Lichtenberg M, Del Giudice C, Sauguet A, Diaz-Cartelle J, Marx C, Strobel A, Schult I, Scheinert D; RANGER SFA Investigators. 12-Month Results From the First-in-Human Randomized Study of the Ranger Paclitaxel-Coated Balloon for Femoropopliteal Treatment. JACC Cardiovasc Interv. 2018 May 28;11(10):934-941. doi: 10.1016/j.jcin.2018.01.276. Epub 2018 May 2. PMID 29730375
- [Result] Zeller T, Baumgartner I, Scheinert D, Brodmann M, Bosiers M, Micari A, Peeters P, Vermassen F, Landini M, Snead DB, Kent KC, Rocha-Singh KJ; IN.PACT DEEP Trial Investigators. Drug-eluting balloon versus standard balloon angioplasty for infrapopliteal arterial revascularization in critical limb ischemia: 12-month results from the IN.PACT DEEP randomized trial. J Am Coll Cardiol. 2014 Oct 14;64(15):1568-76. doi: 10.1016/j.jacc.2014.06.1198. PMID 25301459
- [Result] Mustapha JA, Brodmann M, Geraghty PJ, Saab F, Settlage RA, Jaff MR; Lutonix BTK Study Investigators. Drug-Coated vs Uncoated Percutaneous Transluminal Angioplasty in Infrapopliteal Arteries: Six-Month Results of the Lutonix BTK Trial. J Invasive Cardiol. 2019 Aug;31(8):205-211. PMID 31368893